CLINICAL TRIAL: NCT07153250
Title: Evaluating the Effects of Self-Guided Interventions for Parents of Young Children With Anxiety
Brief Title: Online Parent Education for Child Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Madelaine R. Abel, PhD, Assistant Professor of Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025P001801
Record Dates: First submitted 2025-08-24; First posted 2025-09-03 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-08

CONDITIONS: Anxiety Disorders
Keywords: Anxiety; Parenting; Online Intervention; Child Mental Health
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized (1:1:1 allocation ratio) to receive a three-session program with videos and a workbook or one of two single-session programs with activities. One of the three programs is considered a control condition, but all are education. All parents will repeat baseline evaluation measures 1- and 4-months post baseline. Those in the active groups will also repeat measures at 8-months. Those initially randomized to the control program can be re-randomized after 4 months to either of the active program and will complete subsequent 1- and 4-month follow-up measures post re-randomization.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Project Empower (Experimental): This program is a web-based, self-administered program for parents that takes about 20 minutes to complete. The program includes 5 elements based on the components of cognitive-behavioral therapy.
  Interventions: Behavioral: Project EMPOWER
- Being Brave (Experimental): This program is an online, self-guided program which consists of three brief video-recorded lessons (approximately 20 minutes each) with accompanying knowledge checks and workbook on implementing parent-directed cognitive-behavioral therapy.
  Interventions: Behavioral: Being Brave Parent Education
- Sharing Feelings (Sham Comparator): This program is an online, self-guided 20-minute program, that teaches parents about the importance of sharing feelings and about helpful versus unhelpful expression of emotion.
  Interventions: Behavioral: Sharing Feelings

INTERVENTIONS:
Behavioral: Project EMPOWER — Project EMPOWER is a web-based, self-administered program for parents that takes about 20 minutes to complete.
  Arms: Project Empower
Behavioral: Being Brave Parent Education — Being Brave Parent Education is an online, self-guided program which consists of three brief video-recorded lessons (approximately 20 minutes each) with accompanying knowledge checks and workbook on implementing parent-directed cognitive-behavioral therapy.
  Arms: Being Brave
Behavioral: Sharing Feelings — A self-guided 20-minute educational control, that teaches parents about the importance of sharing feelings and about helpful versus unhelpful expression of emotion.
  Arms: Sharing Feelings

SUMMARY:
The investigators are doing this research to test whether parents of children ages 2-7 can better manage their child's anxiety by completing a brief, online, self-guided parent education program. One way to provide anxiety management skills to more children, and to potentially prevent worsening outcomes, is to offer online and self-guided educational programs that parents can complete without a clinician. This randomized trial will evaluate the effects of two brief, online, self-guided parent education programs designed to improve parents' understanding of anxiety and teach parents way to help their children cope with anxiety. Parents will be randomly assigned to one of the three programs. The main aim of the study is to examine whether the parent programs, compared to an educational control reduce parental accommodation of anxiety across a 1-, 4-, and 8-month follow-up period. As a secondary aim, the investigators will explore whether the parent programs reduce children's anxiety symptoms over the 8-month follow-up period. Results will inform the development of a scalable, low-cost model for promoting access to evidence-based treatment to young children.

DETAILED DESCRIPTION:
Anxiety disorders are very common in children, affecting as many as 30% by adolescence. Even 10% of preschool-age children are already affected. These disorders cause distress and can interfere with academic, social, and family functioning. There are very effective treatments for anxiety disorders, but, on average, kids suffer for four years between onset of their anxiety symptoms and proper diagnosis and treatment. Young children often do not receive treatment because pediatricians, parents, and teachers do not realize that treatment can benefit them and because there is a shortage of providers trained to provide mental health care to young children. Given the importance of early intervention, the investigators are interested in whether parents can learn to better manage their child's anxiety by completing a brief, online, and self-guided parent education program.

Parents will be randomized to one of three self-guided education programs: A three-session program with videos and a workbook and two single-session programs with activities. The programs teach parents how to promote brave behaviors in their child (rather than allowing the child to avoid situations that make them nervous). One of the three programs is considered a control condition, but all are education, and parents will not know whether they are in the control condition until after the 4-month evaluation when they will have the chance to be reassigned to one of the other conditions. The investigators predict that parents who receive one of the active programs, compared to the control, will report greater reductions in parental accommodation across 1-, 4-, and 8-month follow-up. As a secondary hypothesis, the investigators predict that children of parents who receive an active program will show improvements in anxiety symptoms across the 8 month study period.

Because the intervention strategies proposed are brief and easy-to-use, they could be easily implemented as part of routine practice, in much the same way as early intervention for other common childhood health conditions.

ELIGIBILITY:
Inclusion Criteria:

Parents will be eligible to participate if:

1. Their child is between the age of 2 and 7 years-old
2. Their child scores in the elevated range on an age-approrpiate anxiety screening measure
3. Parents are English-speaking
4. Parents are over the age of 18 years old

Exclusion Criteria:

Parents will be excluded if:

(1) Their child shows symptoms of suicidal or homicidal ideation, psychosis, or primary severe mood or behavior disorder (i.e., if treatment for another disorder other than anxiety is indicate prior to treatment for anxiety)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in Pediatric Accommodation Scale, Parent-Report | Change over 8-month follow-up (Baseline to 1-month, 4-month, and 8-month follow-up)
  The Pediatric Accommodation Scale is a parent-report of accommodation of their offspring's anxiety. Parents are asked to rate, on a 5-point scale from 0 (never) to 5 (always), the extent to which they accommodate their child's anxiety or avoidance behaviors. Total scores range from 0 to 25, with higher scores reflecting greater parental accommodation. Parents will report on their accommodation behaviors at baseline , 1-, 4-, and 8-months.

SECONDARY OUTCOMES:
Change in Child Anxiety Symptoms, Parent-Report Total T-Score | Change over 8-month follow-up (Baseline to 1-month, 4-month, and 8-month follow-up)
  To assess child anxiety symptoms, parents will complete either the Spence Child Anxiety Scale (SCAS-P) for children ages 6-7, the Spence Preschool Anxiety Scale (SPAS) for children ages 3-5, or the Infant-Toddler Social and Emotional Assessment Scale (ITSEA) for children aged 2. Each measure produces a Total Anxiety T-Score, which will be used as the secondary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No